CLINICAL TRIAL: NCT05691582
Title: Tolerability of the Immersive Virtual Reality System Grail in Subjects Affected by Rett Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Collaborators: Associazione Italiana Rett (AIRett) O.n.l.u.s. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 885
Record Dates: First submitted 2022-05-26; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Rett Syndrome
Keywords: Virtual Reality; Rett Syndrome; walk
MeSH Terms: conditions — Rett Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): All the subjects recruited have 4 access to GRAIL, in 4 different day, to test their tolerability to the proposals
  Interventions: Device: GRAIL

INTERVENTIONS:
Device: GRAIL — The subjects experiment GRAIL virtual reality for three days, during which they deal with 4 different activities.
  In the first activity subjects are required to ask over the treadmill in a snow environment.
  in the second they are required to stand over the moving platform in a simulation of a boat pitch.
  in the third they have to walk over a bridge with a slope. in the fourth the subjects are required to try so interact with virtual reality and to ski between snowman.
  if it is possible, on the last day a gait analysis is executed

SUMMARY:
The main goal of this study is to investigate the tolerability to the use of the GRAIL system in subjects affected by Rett syndrome, particularly referred to:

1. Grail environment (training in dark conditions, interaction with wide and surrounding screen, positioning over the treadmill);
2. time to prepare a set of body marker in order to execute a gait analysis;
3. walking activity over treadmill, with immersive virtual reality;
4. proprioceptive stimulatione provided by the GRAIL platform;
5. cognitive-attentive span time to the activity proposed. The secondary goal is to understand if a training that avail of treadmill and virtual reality would be useful in the future in improving gait characteristics in subjects affected by Rett syndrome

ELIGIBILITY:
Inclusion Criteria:

* subjects affected by Rett Syndrome that are able to walk with hands support (corresponding to a score ranging from 1 to 3 in item 8 of Rett Syndrome Gross Motor Scale)

Exclusion Criteria:

* subjects unable to walk and with a complete incapacity to undestand verbal directions

Ages: 6 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Rett Syndrome is an X chromosome-associated pathology that reveal almost exclusively in female subjects
Enrollment: 9 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Total score on the Suitability Evaluation Questionnaire (SEQ) | immediately after the treatment
  it is a subjective questionnaire assessing the suitability of the intervention. This is not a health outcome. Indeed SEQ is a questionnaire designed for virtual reality, composed by 13 questions, with a response graded on a 5-point Likert Scale, and a last open question.
  It measures measures enjoyment, sense of being in the system, feeling of success and control, realism, easy-to-understand instructions and general discomfort; furthermore it is aimed to detect issues frequently associated with virtual rehabilitation systems, like dizziness or nausea symptoms, eye discomfort, disorientation or confusion symptoms and sense of progress in rehabilitation. Finally, it evaluates the perceived difficulty of the task and the observed difficulty related with the physical interface used in the system.

SECONDARY OUTCOMES:
Gait analysis spatial parameters: temporal parameters in seconds and kinematics in degrees | immediately after the treatment
  The gait analysis assessment is conducted over the GRAIL (Gait Real-time Analysis Interactive Lab) system .
  It is a laboratory suitable for motion analysis and VR-based rehabilitation. It is composed by a treadmill, provided with two belts that can be driven at different speeds and it is equipped with integrated force platforms. An immersive semicircular screen is placed in front of the treadmill, where VR environments, synchronized with the treadmill movement, are projected. The system uses a Vi-con motion capture system and 3 video cameras to perform motion detection and gait analysis: accordingly, 25 markers were placed on specific anatomical landmarks of the body. Each participant performed a ten-minute familiarization phase and then about 40 steps were acquired.
  Spatiotemporal parameters, such as walking velocity, stance duration, stride length and step width, and kinematic parameters of pelvis, hip, knee and ankle were computed.
Happiness index | immediately after the treatment
  The parameter comes from a taxonomy based on the analysis of the communication of subjects with profound intellectual disabilities. it consists of 12 categories, and each can receive the score "1" when present or "0" when absent

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS E. Medea, Bosisio Parini, Lecco, Italy